CLINICAL TRIAL: NCT07283939
Title: PAGODA: Randomized Trial of a Proactive Graduated Dose Modification Algorithm for FOLFOX Chemotherapy to Prevent Unplanned Delays
Brief Title: Studying the PAGODA Algorithm for Chemotherapy Dose Changes to Prevent Unplanned Treatment Delays
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: A232402CD
Record Dates: First submitted 2025-12-01; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Ampulla of Vater Carcinoma; Appendix Carcinoma; Carcinoma of Unknown Primary With Gastrointestinal Profile; Colon Carcinoma; Esophageal Carcinoma; Gastric Carcinoma; Gastroesophageal Junction Carcinoma; Malignant Digestive System Neoplasm; Rectal Carcinoma; Small Intestinal Carcinoma
MeSH Terms: conditions — Appendiceal Neoplasms; Colonic Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Gastrointestinal Neoplasms; Rectal Neoplasms | interventions — Oxaliplatin; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm B- PAGODA Algorithm (Experimental): Patients receive chemotherapy delays and dose modifications based on PAGODA algorithm followed by treating clinician decision during cycles 2-7 of SOC FOLFOX chemotherapy on study.
  Interventions: Other: PAGODA algorithm; Drug: Oxaliplatin; Drug: Folinic Acid; Drug: Fluorouracil
- Arm A- Physician Discretion (Active Comparator): Patients receive chemotherapy delays and dose modifications at the discretion of the treating clinician during cycles 2-7 of SOC FOLFOX chemotherapy on study.
  Interventions: Drug: Oxaliplatin; Drug: Folinic Acid; Drug: Fluorouracil

INTERVENTIONS:
Other: PAGODA algorithm — use PAGODA algorithm to determine chemotherapy delays and dose modifications
  Arms: Arm B- PAGODA Algorithm
Drug: Oxaliplatin — Given IV
Drug: Folinic Acid — Given IV
  Other Names: Leucovorin
Drug: Fluorouracil — Given IV
  Other Names: 5-FU

SUMMARY:
This study seeks to learn whether using the PAGODA algorithm to guide chemotherapy dosing will lower the chance of unplanned delays during chemotherapy for cancer in the gastrointestinal system compared to usual care.

DETAILED DESCRIPTION:
The primary and secondary objectives of the study:

PRIMARY OBJECTIVE:

I. To compare the proportion of chemotherapy cycles with unplanned delays in patients receiving FOLFOX chemotherapy under standardized usual care (control) versus (vs) according to the PAGODA dose modification algorithm (intervention).

SECONDARY OBJECTIVES:

I. To compare the mean number of health care contact days (time toxicity) for patients receiving FOLFOX chemotherapy according to assignment to the control vs intervention arms.

II. To compare the incidence moderate-to-severe neutropenia (absolute neutrophil count less than 1000/mm3 in patients receiving FOLFOX chemotherapy according to assignment to the control vs intervention arms.

III. To compare the relative dose-intensity of bolus 5-FU, oxaliplatin, and infusional 5-FU in patients receiving FOLFOX chemotherapy according to assignment to the control vs intervention arms, both overall and among the subgroup of participants treated with curative intent.

OUTLINE: This is an interventional study. Patients are randomized to 1 of 2 arms.

ARM A: Patients receive chemotherapy delays and dose modifications at the discretion of the treating clinician during cycles 2-7 of SOC FOLFOX chemotherapy on study.

ARM B: Patients receive chemotherapy delays and dose modifications based on PAGODA algorithm followed by treating clinician decision during cycles 2-7 of SOC FOLFOX chemotherapy on study.

ELIGIBILITY:
Inclusion Criteria:

* * REGISTRATION ELIGIBILITY CRITERIA (STEP 1)

  * Histologic confirmation of invasive cancer that is confirmed or suspected to arise from the gastrointestinal (GI) tract
  * Any stage for which FOLFOX-based chemotherapy is a clinically-indicated, standard-of-care treatment (adjuvant, neoadjuvant, or first-line chemotherapy)
  * Eligible primary tumor sites include the esophagus, gastroesophageal junction, stomach, small intestine, ampulla of Vater, appendix, colon, rectum, and cancers of unknown primary with suspected GI origin
  * Prior systemic therapy for GI cancer (other than cycle 1 of FOLFOX-based chemotherapy) is not allowed. Prior radiation-sensitizing chemotherapy is permitted
  * The planned duration of FOLFOX-based chemotherapy must be at least four cycles (1 cycle = 14 days)
  * Cycle 1, day 1 of FOLFOX-based chemotherapy must be completed 1 to 8 days prior to registration
  * Cycle 1, day 1 of FOLFOX-based chemotherapy must include minimum ordered doses of oxaliplatin (≥ 65 mg/m^2) and infusional 5-FU (2400 mg/m^2/46 hours). Use of the 5-FU bolus is at the discretion of the treating physician
  * Patients who require primary prophylactic white blood cell growth factor with cycle 1 of FOLFOX chemotherapy due to high risk for fever and neutropenia are not eligible
  * History of hypersensitivity reaction to oxaliplatin or other platinum-based drugs, to fluorouracil, or to leucovorin, and the excipients in their formulations are not eligible
  * Age ≥ 18 years
  * ECOG performance status ≤ 2
  * Absolute neutrophil count (ANC) ≥ 1,000/mm^3
  * Platelet count ≥ 100,000/mm^3
  * Total bilirubin ≤ 3 x upper limit of normal (ULN)
  * AST (SGOT)/ALT (SGPT) ≤ 5 x upper limit of normal (ULN)
  * Calc. creatinine clearance ≥ 30 mL/min
  * Not pregnant and not nursing, because this study involves agents that have known genotoxic, mutagenic and teratogenic effects. Therefore, for women of childbearing potential only, a negative pregnancy test done ≤ 30 days prior to registration is required
  * Patients with treated brain metastases are eligible if follow-up brain imaging after CNS-directed therapy shows no evidence of progression
  * Patients with known HIV infection are eligible if receiving effective anti-retroviral therapy with undetectable viral load within 6 months prior to registration
  * Patients with known chronic hepatitis B virus (HBV) infection are eligible if HBV DNA is undetectable when measured within 6 months prior to registration
  * Patients with a known history of hepatitis C virus (HCV) infection are eligible if HCV RNA is undetectable when measured at least 12 weeks after completion of antiviral therapy
  * Patients with known history or current symptoms of cardiac disease are eligible if the New York Heart Association Functional Classification is class I or II
  * Patients with a known history of congenital long QT syndrome are ineligible
  * Patients with known DPD deficiency are ineligible
* * NON-PATIENT (ONCOLOGY PHYSICIAN OR ONCOLOGY ADVANCED PRACTICE PROVIDER ELIGIBILITY:

  * The non-patient provider participant is a medical oncologist or oncology advanced practice provider with responsibility for signing and making necessary modifications to chemotherapy orders for a subject assigned to the intervention arm (Arm B). Non-patient participants may not be enrolled more than once over the course of the study
  * The non-patient participant must be proficient in the English language
  * The non-patient participant must be age 21 years or older

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2030-05-01 (Estimated); Study Completion 2030-05-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of unplanned chemotherapy delays | From cycle 2 to 7 (Undelayed cycle length= 14 days)
  Will employ a generalized linear mixed effects model with logit link function, with a random patient effect to account for clustering of cycles within patients. Will test if additional random effects are needed (e.g., provider or clinic level). Statistical significance will be assessed at the 5% level. Delays will be assessed over cycles 2 through 7, and a delay will be defined as an interval of > 18 days since day 1 of the previous cycle. An unplanned delay will be defined as any delay that was not prospectively planned by day 3 of the previous cycle.

SECONDARY OUTCOMES:
Time toxicity | From registration to 120 days after registration.
  Will use health care contact days as a patient-level measure of time toxicity, as previously described by Gupta et al. Health care contact days will be assessed from electronic health record (EHR) data by recording the number of unique days on which the participant has any in-person contact with the health care system (e.g. for an office visit, chemotherapy treatment, laboratory study, emergency department visit, or other health care service). The mean number of health care contact days will be summarized and compared between the intervention arms using an independent two-sample t-test or Wilcoxon rank sum test. To adjust for multiple comparisons, statistical significance will be evaluated at the 1.25% alpha level.
Moderate-to-severe neutropenia | From the start of cycle 2 to 30 days after start of cycle 7 (undelayed cycle length= 14 days)
  We will assess the patient-level occurrence of ANC less than 1000/mm3 through 30 days after day 1 of the last cycle of protocol treatment. The proportion of patients experiencing ANC less than 1000/mm3 will be summarized and compared between the intervention arms using a Chi-square test for independence or Fisher's Exact test.
Chemotherapy relative dose intensity | Time Frame: From the start of cycle 1 to day 14 of cycle 6 (undelayed cycle length= 14 days).
  Relative dose intensity (RDI) will be individually calculated for 5-FU bolus, oxaliplatin, and infusional 5-FU at the patient-level as the ratio of the delivered dose intensity (dose delivered divided by days elapsed between cycle 1 day 1 and cycle 6 day 14) and the standard dose intensity (standard dose divided by standard treatment interval). The RDI will be summarized and compared between the intervention arms using an independent two-sample t-test or Wilcoxon rank sum test. To adjust for multiple comparisons, statistical significance will be evaluated at the 1.25% alpha level. RDI will be calculated for the entire sample and within treatment intent. For subgroup analyses, statistical significance will be assessed at the 5% level and any positive findings will be considered hypothesis-generating.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel A. Brooks, MD, MPH, Study Chair — Alliance for Clinical Trials in Oncology

IPD SHARING:
Plan to Share IPD: Undecided